CLINICAL TRIAL: NCT02738281
Title: Rett Syndrome, MECP2 Duplication Disorder, and Rett- Related Disorders Natural History Protocol
Brief Title: Natural History of Rett Syndrome & Related Disorders
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Rare Diseases Clinical Research Network (Network); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Alan Percy, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: RDCRN 5211
Record Dates: First submitted 2015-11-22; First posted 2016-04-14 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Rett Syndrome; MECP2 Duplication dIsorder; CDKL5 Disorder; FOXG1 Syndrome
MeSH Terms: conditions — Rett Syndrome; CDKL5 deficiency disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Rett Syndrome: This is a prospective natural history study examining the phenotypic variations of individuals with mutations in MECP2 or meeting the diagnostic criteria for classic (typical) or variant (atypical) Rett syndrome. The overwhelming majority will be female, but males meeting diagnostic criteria will be included. No interventions are planned.
- MECP2 Duplication: This is a prospective natural history study examining the phenotypic variations of individuals with MECP2 duplications. The majority are expected to be males, but females expressing a duplication will be included. No interventions are planned.
- RTT related disorders: This is a prospective natural history study examining individuals, both females and males who do not meet criteria for Rett syndrome, but have a mutation in MECP2, CDKL5, or FOXG1. No interventions are planned.

SUMMARY:
The purpose of this study is to advance understanding of the natural history of Rett syndrome (RTT), MECP2-duplication disorder (MECP2 Dup), CDKL5, FOXG1, and individuals with MECP2 mutations who do not have RTT including the range of clinical involvement and to correlate genotype-phenotype over a broad spectrum of phenotypes. While much has been learned about RTT, improvements are required in understanding the role of factors such as X chromosome inactivation, genetic background, and others including the environment, on the great variability observed even between individuals with the same MECP2 mutation. These data will be essential to the development and conduct of clinical trials that are anticipated from ongoing studies in animal models for RTT. This study will not include clinical trials, but should set the stage for such trials and other translational research projects (e.g., development of biomarkers).

DETAILED DESCRIPTION:
At the present time, effective treatments for RTT, MECP2 Dup, or Rett-related disorders are lacking. Substantial progress has been made in RTT over the past eleven years such that this study represents a narrowing of focus to mutations or duplications of the MECP2 gene and related disorders, including those with phenotypic overlap. Understanding of RTT has advanced remarkably well through the Rett Syndrome Natural History Clinical Protocol (NHS) and correspondingly advancement in the basic science realm has moved forward with equivalent success. Thus, progress in clinical and basic science has led to the establishment of clinical trials and other translational studies that hold promise for additional clinical trials in future. In the process, however, additional MECP2- and RTT-related disorders that were unknown at the time the original proposal have been identified. In addition, substantial clinical variability in individuals with RTT that cannot be explained by differences in mutations alone must be explored further. In fact, variability among individuals with identical mutations has led to the search for additional explanations. At the time of the initial application (2002), just three years after the identification of the gene, MECP2, as the molecular link to RTT, the variation in clinical disorders related to MECP2 mutations or to the related but quite different MECP2 Dup were unknown. Each disorder is characterized by significant neurodevelopmental features related either to alterations in the MECP2 gene or related to phenotypes closely resembling those seen in individuals with RTT. Further, the phenotypic overlap with RTT due to mutations in CDKL5 and FOXG1 was also unexplored. This new study will build on the substantial progress made in understanding both classic and variant RTT and to add these related disorders, MECP2 Dup and the Rett-related disorders including CDKL5, FOXG1, and individuals with MECP2 mutations who do not have RTT. A comprehensive clinical research program will be performed including clinical, neurophysiologic, and molecular and biochemical markers across these different, but related disorders. This protocol will address the natural history components only and will serve as the basis for other study protocols including the neurophysiologic and biomarker studies. Thereby, these studies will represent a continuing pathway to focus and inform not only the ongoing but also the emerging clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both genders and of all ages, with RTT, MECP2 Dup, and, RTT-related disorders including those with mutations or deletions in CDKL5 and FOXG1 genes, or those with RTT (atypical or typical) who are mutation negative.

Exclusion Criteria:

* Individuals who do not meet the above criteria will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Females and males of all ages must have complete testing for MECP2, FOXG1 and CDKL5 genes mutations AND must meet these requirements:
  Gene positive for a sequence mutation, duplication or deletion in one of these 3 genes.
  OR Meet consensus criteria for Rett syndrome (typical or atypical)
Sampling Method: Probability Sample
Enrollment: 1044 (Actual)
Dates: Start 2015-11; Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Clinical longitudinal assessments in Rett syndrome (RTT) as measured by mean growth over 5 years. | at 5 years after enrollment
  subject's height will be measured in inches at baseline and at 5 years. The change will be calculated and then the mean change will be reported.
Clinical and neurobehavioral longitudinal assessments in Rett syndrome (RTT) as measured by mean change in head circumference over 5 years | at 5 years after enrollment
  the mean change in head circumference (measured in Centimeters) will be reported
Clinical and neurobehavioral longitudinal assessments in Rett syndrome (RTT) as measured by mean number of stereotypic movements at 5 years | at 5 years after enrollment
  The mean number of stereotypic movements in a 24 hour period at 5 years.
Clinical and neurobehavioral longitudinal assessments in Rett syndrome (RTT) as the percent of subjects with reported epilepsy at 5 years | 5 years after enrollment
  The Percent of subjects reporting epilepsy by 5 years
Clinical and neurobehavioral longitudinal assessments in Rett syndrome (RTT) as the percent of subjects with reported scoliosis at 5 years | at 5 years after enrollment
  Percent of subjects with reported scoliosis
Clinical and neurobehavioral longitudinal assessments in Rett syndrome (RTT) as the percent of subjects with MECP2 mutations at 5 years | at 5 years after enrollment
  % of subjects with MECP2 mutations to 5 years
Clinical and neurobehavioral longitudinal assessments in Rett syndrome (RTT) as reported by the mean Clinical Severity Scale (CSS) at 5 years | at 5 years after enrollment
  The CSS is the clinical severity scale.
Clinical and neurobehavioral longitudinal assessments in Rett syndrome (RTT) as measured by the mean Motor Behavioral Assessment (MBA) at 5 years | at 5 years after enrollment
  the MBA is the motor behavioral (performance) score
Clinical and neurobehavioral longitudinal assessments in MECP2 duplication syndrome: mean growth rate over 5 years with subjects having MECP2 duplication syndrome | at 5 years after enrollment
  subject's height will be measured in inches at baseline and at 5 years. The change will be calculated and then the mean change will be reported.
Clinical and neurobehavioral longitudinal assessments in MECP2 duplication syndrome: mean change in head circumference 5 years with subjects having MECP2 duplication syndrome | at 5 years after enrollment
  the mean change in head circumference (measured in Centimeters) will be reported
Clinical and neurobehavioral longitudinal assessments in MECP2 duplication syndrome: mean number of stereotypic movements in a 24 hour period at 5 years with subjects having MECP2 duplication syndrome | at 5 years after enrollment
  The mean number of stereotypic movements in a 24 hour period at 5 years.
Clinical and neurobehavioral longitudinal assessments in MECP2 duplication syndrome: percent of subjects reporting scoliosis 5 years with subjects having MECP2 duplication syndrome | at 5 years after enrollment
  Percent of subjects with reported scoliosis
Clinical and neurobehavioral longitudinal assessments in MECP2 duplication syndrome: percent of subjects surviving at 5 years with subjects having MECP2 duplication syndrome | at 5 years after enrollment
  Percent of subjects surviving at 5 years after start of study
Clinical and neurobehavioral longitudinal assessments in MECP2 duplication syndrome: the mean CSS score at 5 years with subjects having MECP2 duplication syndrome | at 5 years after enrollment
  the CSS........
Clinical and neurobehavioral longitudinal assessments in MECP2 duplication syndrome: the mean MAB score at 5 years with subjects having MECP2 duplication syndrome | at 5 years after enrollment
  the MBA........

SECONDARY OUTCOMES:
Quality of Life Measures in RTT | at 5 years post enrollment
  Summative data are provided by the quality of life assessments for children (CHQ), the mean score will.be reported
Quality of Life Measures in MECP2 duplication syndrome | at 5 years post enrollment
  Summative data are provided by the quality of life assessments for children (CHQ), the mean scores will be reported.
Quality of Life Measures in RTT-related disorders. | at 5 years post enrollment
  Summative data are provided by the quality of life assessments for children (CHQ), the mean score will be reported.
Quality of Life Measures in RTT | at 5 years post enrollment
  Summative data are provided by the quality of life assessments from the principal caregiver (SF-36), the mean score will be reported.
Quality of Life Measures in MECP2 duplication syndrome | at 5 years post enrollment
  Summative data are provided by the quality of life assessments from the principal caregiver (SF-36), the mean score will be reported.
Quality of Life Measures in RTT-related disorders | at 5 years post enrollment
  Summative data are provided by the quality of life assessments from the principal caregiver (SF-36), the mean score will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Alan K Percy, MD, Principal Investigator — University of Alabama at Birmingham; Jeffrey L Neul, MD, PhD, Study Director — Vanderbilt University
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCSF Oakland Benioff Children's Hospital, Oakland, California
  - University of California San Diego, San Diego, California
  - University of Colorado Denver, Denver, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Washington University School of Medicine and St. Louis Children's Hospital, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
This consortium will follow the RDCRN agreement to share data. This plan releases data five years after acquisition.

REFERENCES:
- [Background] Hagberg B, Aicardi J, Dias K, Ramos O. A progressive syndrome of autism, dementia, ataxia, and loss of purposeful hand use in girls: Rett's syndrome: report of 35 cases. Ann Neurol. 1983 Oct;14(4):471-9. doi: 10.1002/ana.410140412. PMID 6638958
- [Background] Neul JL, Kaufmann WE, Glaze DG, Christodoulou J, Clarke AJ, Bahi-Buisson N, Leonard H, Bailey ME, Schanen NC, Zappella M, Renieri A, Huppke P, Percy AK; RettSearch Consortium. Rett syndrome: revised diagnostic criteria and nomenclature. Ann Neurol. 2010 Dec;68(6):944-50. doi: 10.1002/ana.22124. PMID 21154482
- [Background] Nan X, Bird A. The biological functions of the methyl-CpG-binding protein MeCP2 and its implication in Rett syndrome. Brain Dev. 2001 Dec;23 Suppl 1:S32-7. doi: 10.1016/s0387-7604(01)00333-3. PMID 11738839
- [Background] Amir RE, Van den Veyver IB, Wan M, Tran CQ, Francke U, Zoghbi HY. Rett syndrome is caused by mutations in X-linked MECP2, encoding methyl-CpG-binding protein 2. Nat Genet. 1999 Oct;23(2):185-8. doi: 10.1038/13810. PMID 10508514
- [Background] Wan M, Lee SS, Zhang X, Houwink-Manville I, Song HR, Amir RE, Budden S, Naidu S, Pereira JL, Lo IF, Zoghbi HY, Schanen NC, Francke U. Rett syndrome and beyond: recurrent spontaneous and familial MECP2 mutations at CpG hotspots. Am J Hum Genet. 1999 Dec;65(6):1520-9. doi: 10.1086/302690. PMID 10577905
- [Background] Suter B, Treadwell-Deering D, Zoghbi HY, Glaze DG, Neul JL. Brief report: MECP2 mutations in people without Rett syndrome. J Autism Dev Disord. 2014 Mar;44(3):703-11. doi: 10.1007/s10803-013-1902-z. PMID 23921973
- [Background] Laurvick CL, de Klerk N, Bower C, Christodoulou J, Ravine D, Ellaway C, Williamson S, Leonard H. Rett syndrome in Australia: a review of the epidemiology. J Pediatr. 2006 Mar;148(3):347-52. doi: 10.1016/j.jpeds.2005.10.037. PMID 16615965
- [Background] Kerr AM, Armstrong DD, Prescott RJ, Doyle D, Kearney DL. Rett syndrome: analysis of deaths in the British survey. Eur Child Adolesc Psychiatry. 1997;6 Suppl 1:71-4. PMID 9452925
- [Background] Guy J, Gan J, Selfridge J, Cobb S, Bird A. Reversal of neurological defects in a mouse model of Rett syndrome. Science. 2007 Feb 23;315(5815):1143-7. doi: 10.1126/science.1138389. Epub 2007 Feb 8. PMID 17289941
- [Background] Garg SK, Lioy DT, Cheval H, McGann JC, Bissonnette JM, Murtha MJ, Foust KD, Kaspar BK, Bird A, Mandel G. Systemic delivery of MeCP2 rescues behavioral and cellular deficits in female mouse models of Rett syndrome. J Neurosci. 2013 Aug 21;33(34):13612-20. doi: 10.1523/JNEUROSCI.1854-13.2013. PMID 23966684
- [Background] Chang Q, Khare G, Dani V, Nelson S, Jaenisch R. The disease progression of Mecp2 mutant mice is affected by the level of BDNF expression. Neuron. 2006 Feb 2;49(3):341-8. doi: 10.1016/j.neuron.2005.12.027. PMID 16446138
- [Background] Tropea D, Giacometti E, Wilson NR, Beard C, McCurry C, Fu DD, Flannery R, Jaenisch R, Sur M. Partial reversal of Rett Syndrome-like symptoms in MeCP2 mutant mice. Proc Natl Acad Sci U S A. 2009 Feb 10;106(6):2029-34. doi: 10.1073/pnas.0812394106. PMID 19208815
- [Background] Archer H, Evans J, Leonard H, Colvin L, Ravine D, Christodoulou J, Williamson S, Charman T, Bailey ME, Sampson J, de Klerk N, Clarke A. Correlation between clinical severity in patients with Rett syndrome with a p.R168X or p.T158M MECP2 mutation, and the direction and degree of skewing of X-chromosome inactivation. J Med Genet. 2007 Feb;44(2):148-52. doi: 10.1136/jmg.2006.045260. Epub 2006 Aug 11. PMID 16905679
- [Background] Leonard H, Bower C. Is the girl with Rett syndrome normal at birth? Dev Med Child Neurol. 1998 Feb;40(2):115-21. PMID 9489500
- [Background] Kerr AM. Early clinical signs in the Rett disorder. Neuropediatrics. 1995 Apr;26(2):67-71. doi: 10.1055/s-2007-979725. PMID 7566455
- [Background] Einspieler C, Kerr AM, Prechtl HF. Abnormal general movements in girls with Rett disorder: the first four months of life. Brain Dev. 2005 Nov;27 Suppl 1:S8-S13. doi: 10.1016/j.braindev.2005.03.014. Epub 2005 Sep 21. PMID 16182501
- [Background] Einspieler C, Kerr AM, Prechtl HF. Is the early development of girls with Rett disorder really normal? Pediatr Res. 2005 May;57(5 Pt 1):696-700. doi: 10.1203/01.PDR.0000155945.94249.0A. Epub 2005 Feb 17. PMID 15718369
- [Background] Downs J, Bebbington A, Kaufmann WE, Leonard H. Longitudinal hand function in Rett syndrome. J Child Neurol. 2011 Mar;26(3):334-40. doi: 10.1177/0883073810381920. Epub 2010 Oct 4. PMID 20921565
- [Background] Downs JA, Bebbington A, Jacoby P, Msall ME, McIlroy O, Fyfe S, Bahi-Buisson N, Kaufmann WE, Leonard H. Gross motor profile in rett syndrome as determined by video analysis. Neuropediatrics. 2008 Aug;39(4):205-10. doi: 10.1055/s-0028-1104575. Epub 2009 Jan 22. PMID 19165708
- [Background] Neul, J.L. Rett Syndrome and MECP2-Related Disorders. in Autism Spectrum Disorders (eds. Amaral, D., Geschwind, D. & Dawson, G.) 776-800 (Oxford University Press, New York, 2011).
- [Background] Nectoux J, Bahi-Buisson N, Guellec I, Coste J, De Roux N, Rosas H, Tardieu M, Chelly J, Bienvenu T. The p.Val66Met polymorphism in the BDNF gene protects against early seizures in Rett syndrome. Neurology. 2008 May 27;70(22 Pt 2):2145-51. doi: 10.1212/01.wnl.0000304086.75913.b2. Epub 2008 Apr 23. PMID 18434641
- [Background] Zeev BB, Bebbington A, Ho G, Leonard H, de Klerk N, Gak E, Vecsler M, Christodoulou J. The common BDNF polymorphism may be a modifier of disease severity in Rett syndrome. Neurology. 2009 Apr 7;72(14):1242-7. doi: 10.1212/01.wnl.0000345664.72220.6a. PMID 19349604
- [Background] Egan MF, Kojima M, Callicott JH, Goldberg TE, Kolachana BS, Bertolino A, Zaitsev E, Gold B, Goldman D, Dean M, Lu B, Weinberger DR. The BDNF val66met polymorphism affects activity-dependent secretion of BDNF and human memory and hippocampal function. Cell. 2003 Jan 24;112(2):257-69. doi: 10.1016/s0092-8674(03)00035-7. PMID 12553913
- [Background] Buchovecky CM, Turley SD, Brown HM, Kyle SM, McDonald JG, Liu B, Pieper AA, Huang W, Katz DM, Russell DW, Shendure J, Justice MJ. A suppressor screen in Mecp2 mutant mice implicates cholesterol metabolism in Rett syndrome. Nat Genet. 2013 Sep;45(9):1013-20. doi: 10.1038/ng.2714. Epub 2013 Jul 28. PMID 23892605
- [Background] Bebbington A, Anderson A, Ravine D, Fyfe S, Pineda M, de Klerk N, Ben-Zeev B, Yatawara N, Percy A, Kaufmann WE, Leonard H. Investigating genotype-phenotype relationships in Rett syndrome using an international data set. Neurology. 2008 Mar 11;70(11):868-75. doi: 10.1212/01.wnl.0000304752.50773.ec. PMID 18332345
- [Background] Ramocki MB, Peters SU, Tavyev YJ, Zhang F, Carvalho CM, Schaaf CP, Richman R, Fang P, Glaze DG, Lupski JR, Zoghbi HY. Autism and other neuropsychiatric symptoms are prevalent in individuals with MeCP2 duplication syndrome. Ann Neurol. 2009 Dec;66(6):771-82. doi: 10.1002/ana.21715. PMID 20035514
- [Background] Peters SU, Hundley RJ, Wilson AK, Carvalho CM, Lupski JR, Ramocki MB. Brief report: regression timing and associated features in MECP2 duplication syndrome. J Autism Dev Disord. 2013 Oct;43(10):2484-90. doi: 10.1007/s10803-013-1796-9. PMID 23456562
- [Background] Friez MJ, Jones JR, Clarkson K, Lubs H, Abuelo D, Bier JA, Pai S, Simensen R, Williams C, Giampietro PF, Schwartz CE, Stevenson RE. Recurrent infections, hypotonia, and mental retardation caused by duplication of MECP2 and adjacent region in Xq28. Pediatrics. 2006 Dec;118(6):e1687-95. doi: 10.1542/peds.2006-0395. Epub 2006 Nov 6. PMID 17088400
- [Background] Van Esch H, Bauters M, Ignatius J, Jansen M, Raynaud M, Hollanders K, Lugtenberg D, Bienvenu T, Jensen LR, Gecz J, Moraine C, Marynen P, Fryns JP, Froyen G. Duplication of the MECP2 region is a frequent cause of severe mental retardation and progressive neurological symptoms in males. Am J Hum Genet. 2005 Sep;77(3):442-53. doi: 10.1086/444549. Epub 2005 Jul 29. PMID 16080119
- [Background] Ramocki MB, Tavyev YJ, Peters SU. The MECP2 duplication syndrome. Am J Med Genet A. 2010 May;152A(5):1079-88. doi: 10.1002/ajmg.a.33184. PMID 20425814
- [Background] Van Esch H. MECP2 Duplication Syndrome. Mol Syndromol. 2012 Apr;2(3-5):128-136. doi: 10.1159/000329580. Epub 2011 Jul 5. PMID 22679399
- [Background] Carvalho CM, Ramocki MB, Pehlivan D, Franco LM, Gonzaga-Jauregui C, Fang P, McCall A, Pivnick EK, Hines-Dowell S, Seaver LH, Friehling L, Lee S, Smith R, Del Gaudio D, Withers M, Liu P, Cheung SW, Belmont JW, Zoghbi HY, Hastings PJ, Lupski JR. Inverted genomic segments and complex triplication rearrangements are mediated by inverted repeats in the human genome. Nat Genet. 2011 Oct 2;43(11):1074-81. doi: 10.1038/ng.944. PMID 21964572
- [Background] Yang T, Ramocki MB, Neul JL, Lu W, Roberts L, Knight J, Ward CS, Zoghbi HY, Kheradmand F, Corry DB. Overexpression of methyl-CpG binding protein 2 impairs T(H)1 responses. Sci Transl Med. 2012 Dec 5;4(163):163ra158. doi: 10.1126/scitranslmed.3004430. PMID 23220634
- [Background] Na ES, Nelson ED, Adachi M, Autry AE, Mahgoub MA, Kavalali ET, Monteggia LM. A mouse model for MeCP2 duplication syndrome: MeCP2 overexpression impairs learning and memory and synaptic transmission. J Neurosci. 2012 Feb 29;32(9):3109-17. doi: 10.1523/JNEUROSCI.6000-11.2012. PMID 22378884
- [Background] Na ES, Nelson ED, Kavalali ET, Monteggia LM. The impact of MeCP2 loss- or gain-of-function on synaptic plasticity. Neuropsychopharmacology. 2013 Jan;38(1):212-9. doi: 10.1038/npp.2012.116. Epub 2012 Jul 11. PMID 22781840
- [Background] Ariani F, Mari F, Pescucci C, Longo I, Bruttini M, Meloni I, Hayek G, Rocchi R, Zappella M, Renieri A. Real-time quantitative PCR as a routine method for screening large rearrangements in Rett syndrome: Report of one case of MECP2 deletion and one case of MECP2 duplication. Hum Mutat. 2004 Aug;24(2):172-7. doi: 10.1002/humu.20065. PMID 15241799
- [Background] Meins M, Lehmann J, Gerresheim F, Herchenbach J, Hagedorn M, Hameister K, Epplen JT. Submicroscopic duplication in Xq28 causes increased expression of the MECP2 gene in a boy with severe mental retardation and features of Rett syndrome. J Med Genet. 2005 Feb;42(2):e12. doi: 10.1136/jmg.2004.023804. No abstract available. PMID 15689435
- [Background] Grasshoff U, Bonin M, Goehring I, Ekici A, Dufke A, Cremer K, Wagner N, Rossier E, Jauch A, Walter M, Bauer C, Bauer P, Horber K, Beck-Woedl S, Wieczorek D. De novo MECP2 duplication in two females with random X-inactivation and moderate mental retardation. Eur J Hum Genet. 2011 May;19(5):507-12. doi: 10.1038/ejhg.2010.226. Epub 2011 Feb 16. PMID 21326285
- [Background] del Gaudio D, Fang P, Scaglia F, Ward PA, Craigen WJ, Glaze DG, Neul JL, Patel A, Lee JA, Irons M, Berry SA, Pursley AA, Grebe TA, Freedenberg D, Martin RA, Hsich GE, Khera JR, Friedman NR, Zoghbi HY, Eng CM, Lupski JR, Beaudet AL, Cheung SW, Roa BB. Increased MECP2 gene copy number as the result of genomic duplication in neurodevelopmentally delayed males. Genet Med. 2006 Dec;8(12):784-92. doi: 10.1097/01.gim.0000250502.28516.3c. PMID 17172942
- [Background] Carvalho CM, Zhang F, Liu P, Patel A, Sahoo T, Bacino CA, Shaw C, Peacock S, Pursley A, Tavyev YJ, Ramocki MB, Nawara M, Obersztyn E, Vianna-Morgante AM, Stankiewicz P, Zoghbi HY, Cheung SW, Lupski JR. Complex rearrangements in patients with duplications of MECP2 can occur by fork stalling and template switching. Hum Mol Genet. 2009 Jun 15;18(12):2188-203. doi: 10.1093/hmg/ddp151. Epub 2009 Mar 26. PMID 19324899
- [Background] Reardon W, Donoghue V, Murphy AM, King MD, Mayne PD, Horn N, Birk Moller L. Progressive cerebellar degenerative changes in the severe mental retardation syndrome caused by duplication of MECP2 and adjacent loci on Xq28. Eur J Pediatr. 2010 Aug;169(8):941-9. doi: 10.1007/s00431-010-1144-4. Epub 2010 Feb 23. PMID 20177701
- [Background] Honda S, Hayashi S, Nakane T, Imoto I, Kurosawa K, Mizuno S, Okamoto N, Kato M, Yoshihashi H, Kubota T, Nakagawa E, Goto Y, Inazawa J. The incidence of hypoplasia of the corpus callosum in patients with dup (X)(q28) involving MECP2 is associated with the location of distal breakpoints. Am J Med Genet A. 2012 Jun;158A(6):1292-303. doi: 10.1002/ajmg.a.35321. Epub 2012 Apr 23. PMID 22528406
- [Background] Vignoli A, Borgatti R, Peron A, Zucca C, Ballarati L, Bonaglia C, Bellini M, Giordano L, Romaniello R, Bedeschi MF, Epifanio R, Russo S, Caselli R, Giardino D, Darra F, La Briola F, Banderali G, Canevini MP. Electroclinical pattern in MECP2 duplication syndrome: eight new reported cases and review of literature. Epilepsia. 2012 Jul;53(7):1146-55. doi: 10.1111/j.1528-1167.2012.03501.x. Epub 2012 May 11. PMID 22578097
- [Background] Lupski JR. Genomic disorders ten years on. Genome Med. 2009 Apr 24;1(4):42. doi: 10.1186/gm42. PMID 19439022
- [Background] Hanashima C, Fernandes M, Hebert JM, Fishell G. The role of Foxg1 and dorsal midline signaling in the generation of Cajal-Retzius subtypes. J Neurosci. 2007 Oct 10;27(41):11103-11. doi: 10.1523/JNEUROSCI.1066-07.2007. PMID 17928452
- [Background] Brancaccio M, Pivetta C, Granzotto M, Filippis C, Mallamaci A. Emx2 and Foxg1 inhibit gliogenesis and promote neuronogenesis. Stem Cells. 2010 Jul;28(7):1206-18. doi: 10.1002/stem.443. PMID 20506244
- [Background] Bahi-Buisson N, Villeneuve N, Caietta E, Jacquette A, Maurey H, Matthijs G, Van Esch H, Delahaye A, Moncla A, Milh M, Zufferey F, Diebold B, Bienvenu T. Recurrent mutations in the CDKL5 gene: genotype-phenotype relationships. Am J Med Genet A. 2012 Jul;158A(7):1612-9. doi: 10.1002/ajmg.a.35401. Epub 2012 Jun 7. PMID 22678952
- [Background] Nemos C, Lambert L, Giuliano F, Doray B, Roubertie A, Goldenberg A, Delobel B, Layet V, N'guyen MA, Saunier A, Verneau F, Jonveaux P, Philippe C. Mutational spectrum of CDKL5 in early-onset encephalopathies: a study of a large collection of French patients and review of the literature. Clin Genet. 2009 Oct;76(4):357-71. doi: 10.1111/j.1399-0004.2009.01194.x. PMID 19793311
- [Background] Brunetti-Pierri N, Paciorkowski AR, Ciccone R, Della Mina E, Bonaglia MC, Borgatti R, Schaaf CP, Sutton VR, Xia Z, Jelluma N, Ruivenkamp C, Bertrand M, de Ravel TJ, Jayakar P, Belli S, Rocchetti K, Pantaleoni C, D'Arrigo S, Hughes J, Cheung SW, Zuffardi O, Stankiewicz P. Duplications of FOXG1 in 14q12 are associated with developmental epilepsy, mental retardation, and severe speech impairment. Eur J Hum Genet. 2011 Jan;19(1):102-7. doi: 10.1038/ejhg.2010.142. Epub 2010 Aug 25. PMID 20736978
- [Background] Wang IT, Allen M, Goffin D, Zhu X, Fairless AH, Brodkin ES, Siegel SJ, Marsh ED, Blendy JA, Zhou Z. Loss of CDKL5 disrupts kinome profile and event-related potentials leading to autistic-like phenotypes in mice. Proc Natl Acad Sci U S A. 2012 Dec 26;109(52):21516-21. doi: 10.1073/pnas.1216988110. Epub 2012 Dec 10. PMID 23236174
- [Background] Huppke P, Held M, Laccone F, Hanefeld F. The spectrum of phenotypes in females with Rett Syndrome. Brain Dev. 2003 Aug;25(5):346-51. doi: 10.1016/s0387-7604(03)00018-4. PMID 12850514
- [Background] Rajaei S, Erlandson A, Kyllerman M, Albage M, Lundstrom I, Karrstedt EL, Hagberg B. Early infantile onset ''congenital'' Rett syndrome variants: Swedish experience through four decades and mutation analysis. J Child Neurol. 2011 Jan;26(1):65-71. doi: 10.1177/0883073810374125. PMID 21212452
- [Background] Nectoux J, Fichou Y, Cagnard N, Bahi-Buisson N, Nusbaum P, Letourneur F, Chelly J, Bienvenu T. Cell cloning-based transcriptome analysis in cyclin-dependent kinase-like 5 mutation patients with severe epileptic encephalopathy. J Mol Med (Berl). 2011 Feb;89(2):193-202. doi: 10.1007/s00109-010-0699-x. Epub 2010 Nov 24. PMID 21107515
- [Background] Ricciardi S, Kilstrup-Nielsen C, Bienvenu T, Jacquette A, Landsberger N, Broccoli V. CDKL5 influences RNA splicing activity by its association to the nuclear speckle molecular machinery. Hum Mol Genet. 2009 Dec 1;18(23):4590-602. doi: 10.1093/hmg/ddp426. Epub 2009 Sep 9. PMID 19740913
- [Background] Weaving LS, Christodoulou J, Williamson SL, Friend KL, McKenzie OL, Archer H, Evans J, Clarke A, Pelka GJ, Tam PP, Watson C, Lahooti H, Ellaway CJ, Bennetts B, Leonard H, Gecz J. Mutations of CDKL5 cause a severe neurodevelopmental disorder with infantile spasms and mental retardation. Am J Hum Genet. 2004 Dec;75(6):1079-93. doi: 10.1086/426462. Epub 2004 Oct 18. PMID 15492925
- [Background] Bahi-Buisson N, Kaminska A, Boddaert N, Rio M, Afenjar A, Gerard M, Giuliano F, Motte J, Heron D, Morel MA, Plouin P, Richelme C, des Portes V, Dulac O, Philippe C, Chiron C, Nabbout R, Bienvenu T. The three stages of epilepsy in patients with CDKL5 mutations. Epilepsia. 2008 Jun;49(6):1027-37. doi: 10.1111/j.1528-1167.2007.01520.x. Epub 2008 Feb 7. PMID 18266744
- [Background] Bahi-Buisson N, Nectoux J, Rosas-Vargas H, Milh M, Boddaert N, Girard B, Cances C, Ville D, Afenjar A, Rio M, Heron D, N'guyen Morel MA, Arzimanoglou A, Philippe C, Jonveaux P, Chelly J, Bienvenu T. Key clinical features to identify girls with CDKL5 mutations. Brain. 2008 Oct;131(Pt 10):2647-61. doi: 10.1093/brain/awn197. Epub 2008 Sep 12. PMID 18790821
- [Background] Fehr S, Wilson M, Downs J, Williams S, Murgia A, Sartori S, Vecchi M, Ho G, Polli R, Psoni S, Bao X, de Klerk N, Leonard H, Christodoulou J. The CDKL5 disorder is an independent clinical entity associated with early-onset encephalopathy. Eur J Hum Genet. 2013 Mar;21(3):266-73. doi: 10.1038/ejhg.2012.156. Epub 2012 Aug 8. PMID 22872100
- [Background] Melani F, Mei D, Pisano T, Savasta S, Franzoni E, Ferrari AR, Marini C, Guerrini R. CDKL5 gene-related epileptic encephalopathy: electroclinical findings in the first year of life. Dev Med Child Neurol. 2011 Apr;53(4):354-60. doi: 10.1111/j.1469-8749.2010.03889.x. Epub 2011 Feb 11. PMID 21309761
- [Background] Elia M, Falco M, Ferri R, Spalletta A, Bottitta M, Calabrese G, Carotenuto M, Musumeci SA, Lo Giudice M, Fichera M. CDKL5 mutations in boys with severe encephalopathy and early-onset intractable epilepsy. Neurology. 2008 Sep 23;71(13):997-9. doi: 10.1212/01.wnl.0000326592.37105.88. PMID 18809835
- [Background] Ward CS, Huang TW, Herrera JA, Samaco RC, Pitcher MR, Herron A, Skinner SA, Kaufmann WE, Glaze DG, Percy AK, Neul JL. Loss of MeCP2 Causes Urological Dysfunction and Contributes to Death by Kidney Failure in Mouse Models of Rett Syndrome. PLoS One. 2016 Nov 9;11(11):e0165550. doi: 10.1371/journal.pone.0165550. eCollection 2016. PMID 27828991
- [Result] Neul JL, Fang P, Barrish J, Lane J, Caeg EB, Smith EO, Zoghbi H, Percy A, Glaze DG. Specific mutations in methyl-CpG-binding protein 2 confer different severity in Rett syndrome. Neurology. 2008 Apr 15;70(16):1313-21. doi: 10.1212/01.wnl.0000291011.54508.aa. Epub 2008 Mar 12. PMID 18337588
- [Result] Kirby RS, Lane JB, Childers J, Skinner SA, Annese F, Barrish JO, Glaze DG, Macleod P, Percy AK. Longevity in Rett syndrome: analysis of the North American Database. J Pediatr. 2010 Jan;156(1):135-138.e1. doi: 10.1016/j.jpeds.2009.07.015. PMID 19772971
- [Result] Tarquinio DC, Motil KJ, Hou W, Lee HS, Glaze DG, Skinner SA, Neul JL, Annese F, McNair L, Barrish JO, Geerts SP, Lane JB, Percy AK. Growth failure and outcome in Rett syndrome: specific growth references. Neurology. 2012 Oct 16;79(16):1653-61. doi: 10.1212/WNL.0b013e31826e9a70. Epub 2012 Oct 3. PMID 23035069
- [Result] Kalman LV, Tarleton JC, Percy AK, Aradhya S, Bale S, Barker SD, Bayrak-Toydemir P, Bridges C, Buller-Burckle AM, Das S, Iyer RK, Vo TD, Zvereff VV, Toji LH. Development of a genomic DNA reference material panel for Rett syndrome (MECP2-related disorders) genetic testing. J Mol Diagn. 2014 Mar;16(2):273-9. doi: 10.1016/j.jmoldx.2013.11.004. Epub 2014 Feb 7. PMID 24508304
- [Result] Cuddapah VA, Pillai RB, Shekar KV, Lane JB, Motil KJ, Skinner SA, Tarquinio DC, Glaze DG, McGwin G, Kaufmann WE, Percy AK, Neul JL, Olsen ML. Methyl-CpG-binding protein 2 (MECP2) mutation type is associated with disease severity in Rett syndrome. J Med Genet. 2014 Mar;51(3):152-8. doi: 10.1136/jmedgenet-2013-102113. Epub 2014 Jan 7. PMID 24399845
- [Result] Neul JL, Lane JB, Lee HS, Geerts S, Barrish JO, Annese F, Baggett LM, Barnes K, Skinner SA, Motil KJ, Glaze DG, Kaufmann WE, Percy AK. Developmental delay in Rett syndrome: data from the natural history study. J Neurodev Disord. 2014;6(1):20. doi: 10.1186/1866-1955-6-20. Epub 2014 Jul 22. PMID 25071871
- [Result] Killian JT, Lane JB, Cutter GR, Skinner SA, Kaufmann WE, Tarquinio DC, Glaze DG, Motil KJ, Neul JL, Percy AK. Pubertal development in Rett syndrome deviates from typical females. Pediatr Neurol. 2014 Dec;51(6):769-75. doi: 10.1016/j.pediatrneurol.2014.08.013. Epub 2014 Aug 29. PMID 25283752
- [Result] Tarquinio DC, Hou W, Neul JL, Lane JB, Barnes KV, O'Leary HM, Bruck NM, Kaufmann WE, Motil KJ, Glaze DG, Skinner SA, Annese F, Baggett L, Barrish JO, Geerts SP, Percy AK. Age of diagnosis in Rett syndrome: patterns of recognition among diagnosticians and risk factors for late diagnosis. Pediatr Neurol. 2015 Jun;52(6):585-91.e2. doi: 10.1016/j.pediatrneurol.2015.02.007. Epub 2015 Feb 16. PMID 25801175
- [Result] Killian JT Jr, Lane JB, Lee HS, Pelham JH, Skinner SA, Kaufmann WE, Glaze DG, Neul JL, Percy AK. Caretaker Quality of Life in Rett Syndrome: Disorder Features and Psychological Predictors. Pediatr Neurol. 2016 May;58:67-74. doi: 10.1016/j.pediatrneurol.2015.12.021. Epub 2016 Jan 11. PMID 26995066
- [Result] Sajan SA, Jhangiani SN, Muzny DM, Gibbs RA, Lupski JR, Glaze DG, Kaufmann WE, Skinner SA, Annese F, Friez MJ, Lane J, Percy AK, Neul JL. Enrichment of mutations in chromatin regulators in people with Rett syndrome lacking mutations in MECP2. Genet Med. 2017 Jan;19(1):13-19. doi: 10.1038/gim.2016.42. Epub 2016 May 12. PMID 27171548
- [Result] Lane JB, Salter AR, Jones NE, Cutter G, Horrigan J, Skinner SA, Kaufmann WE, Glaze DG, Neul JL, Percy AK. Assessment of Caregiver Inventory for Rett Syndrome. J Autism Dev Disord. 2017 Apr;47(4):1102-1112. doi: 10.1007/s10803-017-3034-3. PMID 28132121
- [Result] Tarquinio DC, Hou W, Neul JL, Kaufmann WE, Glaze DG, Motil KJ, Skinner SA, Lee HS, Percy AK. The Changing Face of Survival in Rett Syndrome and MECP2-Related Disorders. Pediatr Neurol. 2015 Nov;53(5):402-11. doi: 10.1016/j.pediatrneurol.2015.06.003. Epub 2015 Jun 26. PMID 26278631
- [Derived] Neul JL, Benke TA, Marsh ED, Suter B, Silveira L, Fu C, Peters SU, Percy AK; Rett syndrome Natural History Study Group. Top caregiver concerns in Rett syndrome and related disorders: data from the US natural history study. J Neurodev Disord. 2023 Oct 13;15(1):33. doi: 10.1186/s11689-023-09502-z. PMID 37833681
- [Derived] Saby JN, Peters SU, Benke TA, Standridge SM, Swanson LC, Lieberman DN, Olson HE, Key AP, Percy AK, Neul JL, Nelson CA, Roberts TPL, Marsh ED. Comparison of evoked potentials across four related developmental encephalopathies. J Neurodev Disord. 2023 Mar 4;15(1):10. doi: 10.1186/s11689-023-09479-9. PMID 36870948
- [Derived] Buchanan CB, Stallworth JL, Joy AE, Dixon RE, Scott AE, Beisang AA, Benke TA, Glaze DG, Haas RH, Heydemann PT, Jones MD, Lane JB, Lieberman DN, Marsh ED, Neul JL, Peters SU, Ryther RC, Skinner SA, Standridge SM, Kaufmann WE, Percy AK. Anxiety-like behavior and anxiolytic treatment in the Rett syndrome natural history study. J Neurodev Disord. 2022 May 14;14(1):31. doi: 10.1186/s11689-022-09432-2. PMID 35568815
- See also: International Rett Syndrome Foundation website — http://www.rettsyndrome.org/